CLINICAL TRIAL: NCT04971447
Title: Effects of Plasma Extracellular Vesicles on Endothelial Function in Transgender Subjects
Brief Title: Extracellular Vesicles and Endothelial Function in Transgender Subjects
Acronym: Evinge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21.03.30.69624
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2021-07

CONDITIONS: Transgenderism
Keywords: transgender persons; hormonal therapy
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group: transgender men (Experimental)
  Interventions: Drug: gender affirming hormonal treatment in transgender men
- Groupe: control cis-gender women (No Intervention)
- Group: transgender women (Experimental)
  Interventions: Drug: gender affirming hormonal treatment in transgender women
- Groupe: control cis-gender men (No Intervention)

INTERVENTIONS:
Drug: gender affirming hormonal treatment in transgender men — testosterone enanthate
  Arms: Group: transgender men
Drug: gender affirming hormonal treatment in transgender women — GnRH agonists + estrogen
  Arms: Group: transgender women

SUMMARY:
Cardiovascular diseases are the leading cause of mortality. In women, the prevalence of cardiovascular diseases is lower and the presentation of coronary events often atypical. The lack of evidence is related in part to the methodology of studies not considering sex as an essential biological variable. Hormonal treatment is prescribed in transgender subjects to promote the development of sexual characteristics of the desired sex. Early cardiovascular effects of hormonal treatment have been reported in transgender men, while long-term mortality is higher in transgender women. The aim of this project is to study the effects of gender affirming hormonal treatment on arterial stiffness in young transgender subjects followed at the University Hospital of Nancy.

ELIGIBILITY:
Inclusion Criteria:

* Trasgender subject demanding gender affirming hormonal therapy

Exclusion Criteria:

* Previous hormonal therapy
* Pregnancy
* Chronic disease
* Cancer
* Obesity
* Drug abuse
* Alcohol
* Tabac

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — yes
Enrollment: 136 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
pulse wave velocity | 24 months
  measurement of arterial stiffness